CLINICAL TRIAL: NCT05053204
Title: Based on the THINC-it Tool to Explore the Characteristics and Related Factors of Cognitive Impairment in the Acute Stage of Unipolar and Bipolar Depression
Brief Title: Influence Factors and Cognitive Characteristics in Unipolar and Bipolar Depression:Based on the THINC-it Tool
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: PWRq2021-59
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2021-09

CONDITIONS: Cognitive Impairments
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- unipolar depression group: In accordance with the diagnostic criteria of ICD-10 Unipolar depressive disorder, outpatients or inpatients in the Department of mood Disorders, Mental Health Center of Pudong New area.
- bipolar depression group: In accordance with the diagnostic criteria of ICD-10 Bipolar depression , outpatients or inpatients in the Department of mood Disorders, Mental Health Center of Pudong New area.
- healthy control group: Any mental disorder that does not meet the diagnosis of ICD-10, and the society recruits healthy controls who match the sex, age and education level of the patients in the case-group.

INTERVENTIONS:
Other:
  Groups: bipolar depression group; unipolar depression group

SUMMARY:
Cognitive impairment is the core symptom of unipolar and bipolar depression, which seriously affects the prognosis of the disease and the rehabilitation of social function. There is no unified conclusion in the field and severity of cognitive impairment, and the cause of cognitive impairment is unknown, which may be related to many factors. In this study,the THINC-it tool was used to study the characteristics of cognitive impairment in unipolar and bipolar depression by longitudinal follow-up, which provides a theoretical basis for the differential diagnosis of unipolar and bipolar depression. Early identification and intervention of risk factors can improve the prognosis of the disease.

DETAILED DESCRIPTION:
there is some cognitive impairment in patients with unipolar and bipolar depression. There is no unified conclusion in the field and severity of cognitive impairment, and the cause of cognitive impairment is unknown, which may be related to many factors. The THINC-it is a simple, fast and free cognitive assessment tool for cognitive impairment screening of unipolar and bipolar depression.

This study includes three steps.

1. baseline: demographic data, theTHINC-it tool , clinical scales（HAMD-17,HAMA、YMRS、PSQI） evaluation and Laboratory examination（blood glucose, blood lipids, BMI）
2. follow-up (4 week): Clinical scales and THINC-it tool were evaluated in unipolar and bipolar depression.
3. follow-up (12 weeks): all patients with bipolar depression were evaluated by clinical scales, THINC-it test.

ELIGIBILITY:
Inclusion Criteria:

Case group:

1、Participants in psychiatric outpatients and inpatients are able and willing to provide informed consent.

2. The participants were male or female aged between 18 and 60, with junior high school education or above.

3. According to ICD-10 criteria, participants were diagnosed with Unipolar and bipolar depressive disorder.

4. The total score of Young's Mania scale ((YMRS)) of the participants was less than 5 and HAMD-17 was greater than17.

5. Subjects received stable mood stabilizers at least two weeks before the study visit, such as SSRIs antidepressants.

6. The combination or use of supportive psychotherapy is allowed.

Control group:

1.it did not meet any of the diagnostic criteria in ICD-10 in the past or at present.

2.18-60 years old, junior high school education or above. 3.Have sufficient audio-visual skills to complete the necessary examinations of the study.

4.Willing to participate in this study, and the informed consent form was signed by the subjects.

Exclusion Criteria:

1. Current alcohol and / or substance use disorders.
2. Any drugs that may affect cognitive function, such as psychotropic stimulants, corticosteroids, and receptor blockers.
3. Benzodiazepines were used within 12 hours and alcohol consumption within 8 hours before using the THINC-it tool.
4. The patients have some serious physical conditions.
5. The patients received electroconvulsive therapy ((ECT)) in the past 6 months.
6. They are serious negative suicidal concepts and behaviors.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: According to the diagnostic criteria of ICD-10 Unipolar and bipolar depressive disorder, 40 patients with Major depressive disorder, 40 patients with bipolar depression and 40 healthy controls matched with the sex, age and education level of the patients in the case group served as healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
the THINC-it Tool | up to 12 week
  The composite THINC-it tool score is the integrated total score of results from performance on five sub-component cognitive tests of the THINC-it tool.

SECONDARY OUTCOMES:
HAMD-17 | up to 12 week
  Assess the state of depression
HAM-A | up to 12 week
  Assessing anxiety state
Pittsburgh Sleep Quality Index，PSQI | up to 12 week
  Evaluate sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, M.D., Ph.D, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center IRB, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided